Statistical Analysis Plan

Study Title: New Options for Treating Knee Osteoarthritis Pain

NCT Number: NCT05541718

Document Date Last Approved: 7/12/2022

Emerald Gate Charitable Trust 07/12/2022 – <u>University of Utah</u> Project Authorization Page 10 of 15

**STATISTICAL APPROACH.** Linear mixed models will evaluate study outcomes by examining the Treatment (BT vs. NHP vs. MM vs. WL) X Time (Primary and Secondary Trait: Baseline vs. 4-week vs. 8-week; Secondary State: Treatment Session 1 vs. 2 vs. 3 vs. 4) interaction. Intention-to-treat and perprotocol analyses will be performed. Structural equation modeling will evaluate whether therapeutic mechanisms statistically mediate study outcomes.